CLINICAL TRIAL: NCT02896842
Title: A Prospective Randomized Phase II Study Evaluating the Monitoring of Imatinib Mesylate (Glivec®) Plasmatic Through Level in Patients Newly Diagnosed With Chronic Phase Chronic Myelogenous Leukaemia (CP-CML).
Brief Title: A Prospective Randomized Phase II Study Evaluating the Monitoring of Imatinib Mesylate Plasmatic Through Level in Patients Newly Diagnosed With CP-CML
Acronym: OPTIMIMATINIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Philippe ROUSSELOT, Study coordonator, Versailles Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/38_ Optim Imatinib
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Arm (No Intervention): cohort 3: Imatinib through dosage ≥ 1000 ng/ml
- Active comparator (Active Comparator): Cohort 2 : Imatinib standard dose Imatinib through dosage < 1000 ng/ml
  Interventions: Other: active comparator
- Experimental arm (Experimental): Cohort 1 : dose adjustment based on trough plasmatic level value Imatinib through dosage < 1000 ng/ml
  Interventions: Drug: Posology dose modification

INTERVENTIONS:
Drug: Posology dose modification
  Other Names: Cohort 1 : dose adjustment based on trough plasmatic
  Arms: Experimental arm
Other: active comparator
  Other Names: Cohort 2 : Imatinib standard dose
  Arms: Active comparator

SUMMARY:
Imatinib mesylate (Gleevec/Glivec, IM) is currently the gold standard or CML-CP front line therapy. The recommended dose of IM is 400 mg/day. The rates of complete cytogenetic responses at 3, 6 and 12 months are 27%, 50% and 69% respectively. The optimal IM daily dose is not yet determined and randomized studies addressing this question are on-going. First results from the TOPS trial (EHA 2008 congress) suggest a more rapid kinetic of response for patients treated with imatinib high dose. Recent studies revealed that initial Imatinib plasmatic dosage is predictive for achieving complete cytogenetic responses (CCR) and that a dosage of 1000 ng/ml is associated with a higher proportion of major molecular responses (MMR) (Picard et al., Blood 2007, Larson et al. Blood 2007).

Results from the study of Larson et al. indicate that around 40% of the patients had a trough plasmatic level below 1000 ng/ml after day 28 of imatinib 400 mg/d. The major molecular response rate at 12 months for the patients with the lower plasmatic through level is 25.4% compared to 40.1% for the patients with a plasmatic dosage over 800 to 1000 ng/ml.

Investigators propose to adapt the imatinib daily dose in case of imatinib through plasmatic level at day 28 below 1000 ng/ml. Patients with a trough plasmatic dosage ≤ 1000 ng/ml will be randomized between a prospective adaptation strategy of the imatinib daily dose (cohort 1) versus observation only (cohort 2). The patients with adequate imatinib dosage (> 1000 ng/ml) will be followed up according the ELN recommendation (cohort 3). Imatinib trough plasmatic level will then be rechecked every month thereafter for patients in cohort 1 and cohort 2 and every three months in cohort 3. The first endpoint of the study will be the rate of major molecular response at 12 months in cohort 1. Our hypothesis is to improve the 12 months MMR rate with the optimized strategy (cohort 1) from 25% of MMR at 12 months to 40% of MMR at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥ 18 years
2. Philadelphia chromosome positive newly diagnosed chronic myelogenous leukaemia (≤ 4 months) in first chronic phase.
3. Not previously treated with tyrosine kinase inhibitors other than imatinib
4. Prior treatment with imatinib during less than 13 weeks
5. Signed written inform consent
6. Women of childbearing potential (WOCBP) must be using an adequate method of contraception

Exclusion Criteria:

1. Patients with BCR-ABL positive, Philadelphia negative CML
2. Patient previously treated with TKI other than imatinib
3. Pregnancy
4. Active malignancy
5. Concurrent severe diseases which exclude the administration of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2010-09; Primary Completion 2015-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The major molecular response rate at 12 months in cohort 1. | 12 months

SECONDARY OUTCOMES:
Complete cytogenetic response at 6 and 12 months | 12 months
Major molecular response rate at 12 months in cohort 2 and cohort 3. | 12 months
Major molecular response at 3, 6, and 9 months | 9 months
Complete molecular response 6 and 12 months | 12 months
Relationship between plasmatic dosage and efficacy | 12 months
Relationship between plasmatic dosage and tolerance | 12 months
Progression free survival | 5 years
Event free survival | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - CHU angers, Angers
  - CH d'Annecy, Annecy
  - CH argenteuil, Argenteuil
  - CHU Bordeaux, Bordeaux
  - Institut Bergonié, Bordeaux
  - CH Boulogne, Boulogne
  - CHU CAEN, Caen
  - CH de Dieppe, Dieppe
  - CH Dunkerque, Dunkirk
  - CH Versailles, Le Chesnay
  - CHU Lille, Lille
  - CHU Lyon, Lyon
  - CH Meaux, Meaux
  - Hopital Bon secours, Metz
  - CHU Nice, Nice
  - Hopital La Source, Orléans La Source
  - Hopital Necker, Paris
  - CHU Rennes, Rennes
  - Hopital Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No